CLINICAL TRIAL: NCT05785819
Title: A Randomized, Double-Blind, Phase 2 Pilot Study of VLX-1005 Versus Placebo in Participants With Suspected Heparin Induced Thrombocytopenia Treated With Background Standard of Care
Brief Title: A Phase 2 Study of VLX-1005 Versus Placebo in Suspected Heparin Induced Thrombocytopenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Veralox Therapeutics Business Decision.
Sponsor: Veralox Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VLX-1005-003
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Thrombocytopenia, Immune; Heparin Induced Thrombocytopenia
Keywords: Heparin; Thrombocytopenia; Platelets
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VLX-1005 (Experimental): VLX-1005 200 mg given every 12 hours by intravenous infusion over 1 hour.
  Interventions: Drug: VLX-1005
- Placebo (Placebo Comparator): Placebo given every 12 hours by intravenous infusion over 1 hour.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VLX-1005 — VLX-1005, a 12-LOX enzyme inhibitor
  Other Names: 12-LOX enzyme inhibitor
  Arms: VLX-1005
Drug: Placebo — Placebo matching VLX-1005
  Other Names: Inactive substance similar in appearance to VLX-1005
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VLX-1005, a 12-lipoxygenase (12-LOX) enzyme inhibitor in treating heparin induced thrombocytopenia (HIT). Participants with suspected HIT will receive the usual standard of care, and will be assigned randomly to either VLX-1005 or placebo treatment. The study will measure important outcomes including platelet count, stroke, pulmonary embolus (clot to the lungs) and bleeding.

DETAILED DESCRIPTION:
Over 12 million patients are treated with heparin each year in the United States. Heparin induced thrombocytopenia (HIT) is a recognized complication of heparin therapy and is characterized by the formation of antibodies to heparin and platelet factor 4 (PF4). The scale of the clinical problem is illustrated by cardiopulmonary bypass patients, half of whom develop antibodies to PF4/heparin complexes. In a significant proportion of such seropositive HIT patients, these antibodies will bind to and activate platelets, resulting in a drop in the number of platelets (thrombocytopenia) and activation of the coagulation (clotting) system. Formation of clots in this manner can lead to stroke, heart attacks, damage to internal organs or to limbs, and even death.

The current standard of care with anticoagulants such as argatroban or bivalirudin have not proven effective in reducing poor outcomes in HIT: major morbidity and death rates remain high (> 20%). In addition, these anticoagulants increase the risk of major bleeding (~20%) which can prove to be a fatal complication of such therapy.

VLX-1005 has been developed to address the major unmet clinical need for safer, more effective therapy for HIT. VLX-1005 is a drug that blocks the 12-lipoxygenase (12-LOX) pathway that is believed to be responsible for platelet activation in HIT. In animal models of HIT, VLX-1005 can prevent or treat HIT and halt the development of both thrombocytopenia and abnormal blood clots. The drug has not been associated with increased bleeding in either animals or healthy human volunteers.

The current study will enroll patients suspected of having HIT by clinical measures (4T score) and by laboratory testing (heparin-PF4 immunoassay). Patients will be randomly assigned in a double-blind fashion to either VLX-1005 intravenously or placebo. All patients will receive current guideline mandated therapy for HIT that will include the standard of care anticoagulation: either argatroban or bivalirudin. Patients will be treated for 7 to 14 days until the platelet count has recovered into the normal range. The study will measure important outcomes including platelet count recovery time, stroke, pulmonary embolus, deep vein thrombosis, myocardial infarction, limb and organ injury, and major bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants ≥ 18 years of age.
2. Able to provide informed consent or have informed consent provided on their behalf by a primary caregiver prior to study-related activities being initiated.
3. Recent unfractionated heparin or low-molecular-weight heparin exposure.
4. Qualifying platelet count < 150 X 10^9/L and clinical 4T score of ≥ 4; candidate for argatroban or bivalirudin treatment.
5. Positive PF4-immunoassay (eg, ELISA [≥ 1.0 optical density units], LIA [≥ 1.0 U/mL], CLIA [≥ 1.0 U/mL]).

   -

Exclusion Criteria:

1. Treatment with argatroban or bivalirudin for ≥ 60 hrs prior to randomization.
2. Following discontinuation of heparin, participants cannot be treated with a non-heparin anti-coagulant for ≥ 60 hours.
3. Current renal dialysis.
4. Pregnant or lactating women.
5. Have participated in any other investigational drug trial within 30 days of dosing or 5 half-lives (whichever is longer) in the current study.
6. In the opinion of the investigator, unlikely to comply with key elements of the protocol or otherwise inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Time to recovery of platelet count to ≥ 150 X 10^9/L in patients with a positive serotonin release assay | Up to 14 days
  Time to platelet count recovery; defined as the time from the first dose of study drug to the time of the first of 2 consecutive platelet count recoveries to ≥ 150 X 10^9/L in patients with positive serotonin release assay (SRA+) confirmed HIT.

SECONDARY OUTCOMES:
Composite of death, amputation, new thrombosis, stroke, systemic embolism, myocardial infarction, deep vein thrombosis or pulmonary embolism, skin necrosis, limb gangrene, organ ischemia or infarction | Up to14 days
  Proportion of participants with incidence of the composite of death, amputation, new thrombosis, stroke, systemic embolism, myocardial infarction, deep vein thrombosis or pulmonary embolism, skin necrosis, limb gangrene, organ ischemia or infarction
Incidence of death, amputation, new thrombosis, stroke, systemic embolism, myocardial infarction, deep vein thrombosis or pulmonary embolism, organ ischemia or infarction | Up to14 days
  Time from study drug initiation to any incidence of the composite of death, amputation, new thrombosis, stroke, systemic embolism, myocardial infarction, deep vein thrombosis or pulmonary embolism, skin necrosis, limb gangrene, organ ischemia or infarction
Time from the first dose of study drug to change to oral anti-coagulant treatment | Up to14 days
  Time from initiation of therapy to switching to oral treatment
Time from study drug initiation to each element of the composite as a separate endpoint: death, amputation, new thrombosis, stroke, systemic embolism, myocardial infarction, deep vein thrombosis or pulmonary embolism, organ ischemia or infarction | Up to14 days
  Measurement of important clinical outcomes by time to event
Proportion of participants with any element of the composite as a separate endpoint: death, amputation, new thrombosis, stroke, systemic embolism, myocardial infarction, deep vein thrombosis or pulmonary embolism, organ ischemia or infarction | Up to14 days
  Measurement of proportion of participants with important clinical outcomes
Time from study drug initiation to occurrence of any incidence of International Society on Thrombosis and Haemostasis (ISTH) major bleeding | Up to14 days
  Incidence of major bleeding by time to event
Proportion of participants with incidence of major bleeding as defined by ISTH criteria | Up to14 days
  Measurement of proportion of participants who develop major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: John Alexander, MD, Study Chair — Duke Clinical Research Institute
Locations (14):
- United States (14):
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Universiy of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Carilion Medical Center, Roanoke, Virginia
  - University of Washington, Seattle, Washington
  - Versiti at Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No